CLINICAL TRIAL: NCT02229578
Title: Lidocaine In The Treatment of Post-operative Pain Management From a Donor Site After Split Thickness Skin Graft Harvesting Following Thermal Injury
Brief Title: Lidocaine For Treatment of Post-operative Pain From Donor Sites Following Burn Injury.
Acronym: LidocaineBurn
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB201400019; OCR18920 (Other: UF OnCore)
Record Dates: First submitted 2014-08-27; First posted 2014-09-01 (Estimated); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Pain
Keywords: Burn pain; lidocaine; donor site pain; Narcotic use
MeSH Terms: conditions — Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine Treatment Group (Experimental): Subjects in this group will receive a nonpyrogenic solution of lidocaine 2% in isotonic saline (Solution A) sprayed on the donor site of the grafted skin prior to emergence from general anesthesia. A total maximum of 7mg/kg of lidocaine solution will be available for administration. Prior to spraying of the Solution A, the donor site will be soaked with epinephrine soaked towels as per routine burn care. The site will then be covered with TheraBond dressing as per standard burn care.
  Interventions: Drug: Lidocaine
- Placebo Treatment Group (Placebo Comparator): Subjects in this group will receive a nonpyrogenic solution of isotonic saline (Solution B) sprayed over the donor site. Prior to spraying of the Solution B, the donor site will be soaked with epinephrine soaked towels as per routine burn care. The site will then be covered with TheraBond dressing as per standard burn care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Subjects in this group will receive a nonpyrogenic solution of lidocaine 2% in isotonic saline (Solution A) sprayed on the donor site of the grafted skin prior to emergence from general anesthesia. A total maximum of 7mg/kg of lidocaine solution will be available for administration. Prior to spraying of the Solution A, the donor site will be soaked with epinephrine soaked towels as per routine burn care. The site will then be covered with TheraBond dressing as per standard burn care.
  Arms: Lidocaine Treatment Group
Drug: Placebo — Subjects in this group will receive a nonpyrogenic solution of isotonic saline (Solution B) sprayed over the donor site. Prior to spraying of the Solution B, the donor site will be soaked with epinephrine soaked towels as per routine burn care. The site will then be covered with TheraBond dressing as per standard burn care.
  Other Names: Saline
  Arms: Placebo Treatment Group

SUMMARY:
Burn pain is known to be one the most severe forms of acute pain often requiring large amounts of narcotics in addition to other adjuvants. Topical lidocaine is effective for controlling pain in various settings including dressing changes of burns. The aim of this study is to demonstrate the effectiveness of topical lidocaine in decreasing pain scores and narcotic requirements when applied to donor graft sites while at the same time not interfering with the standard of care TheraBond dressing. During this study the investiagtors will be monitoring for evidence of delayed wound healing, and surgical site infection.

DETAILED DESCRIPTION:
Pain from burns is a severe form of acute pain that requires aggressive use of opioids. Even with the implementation of multiple modalities for analgesia, pain from skin debridements and grafting procedures remains a challenge to control. Local anesthetics have been used for pain relief in burn patients previously as a topical gel or IV infusion and have been found to significantly reduce medication consumption, without apparent adverse effects on wound healing. Lidocaine actually has potent anti-inflammatory effects which could be advantageous on wounds. In addition, topical application of lidocaine to wounds result in different degrees of systemic absorption. High concentrations of lidocaine have potential for central nervous system (seizures (>5mg/L)) and cardiovascular toxicity (arrhythmias (>9mg/L)). Plasma concentration of lidocaine depend upon drug dose, rate of absorption, patient weight, physical status and thickness of skin harvested. A prior study where up to 6.7mg/kg of 2% lidocaine with epinephrine was sprayed on donor graft sites found that systemic lidocaine levels were far below toxic levels at their peak (average level of 1.4, with maximum level at 2.2). In this study the levels peaked between 30 and 60 minutes and systemic levels of lidocaine were detectable 6 hours following application of the solution. Studies have demonstrated the beneficial effects of systemic lidocaine administered via IV infusions in reducing perioperative pain scores.Topical lidocaine is effective as a topical anesthetic in multiple clinical trials however only two studies to date has shown that topical lidocaine applied to skin-harvest sites produces an analgesic effect, reduces narcotic requirements while not affecting wound healing or causing toxic blood concentrations. In both these studies systemic intravenous lidocaine levels were monitored and were found to be significantly below toxic limits. The use of topical lidocaine on donor sites is still not widely used, partly for fear the lidocaine will interfere with wound healing and/or dressing adherence. No study to date has demonstrated lidocaine solution to be effective on burn sites when used in conjunction with TheraBond silver foam dressing. TheraBond is an absorbent, atraumatic dressing coated with ionic silver that is routinely used on donor sites at the University of Florida. This study will also offer additional supporting evidence that topical lidocaine is effective in post operative pain management of donor skin sites and should be more widely utilized. In addition, this study will serve as a stepping stone for analyzing different local anesthetic solutions in the future and the potential for reapplication to surgical sites.

The purpose of this study is to offer the medical community data on a simple and relatively cheap adjuvant that can be utilized to help reduce the amount of post-operative pain and narcotic requirement in burn patients requiring skin grafts.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have suffered second to third degree burns requiring a single split thickness skin graft surgery.
* Donor sites will be between 3-15% TBSA.

Exclusion Criteria:

* Patients who have history of chronic pain,
* opioid abuse history,
* major renal and/or liver dysfunction,
* history of seizures or major neurologic deficiencies,
* allergy to local anesthetics,
* reported allergy to hydromorphone,
* pregnancy, or
* currently have other injuries that significantly contribute to pain (i.e. multi-trauma patients) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Fahy, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Shands Hospital, University of Florida, Gainesville, Florida
  - Shands Hospital, Gainesville, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine Treatment Group | Placebo Treatment Group
Started | 19 | 15
Completed | 16 | 12
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Treatment Group | Placebo Treatment Group | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (15.1) | 44.1 (14.7) | 43.7 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 15 | 11 | 26
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Pain Change
Description: Improvement of pain perception for those receiving lidocaine vs those that do not. Pain will be measured by the Verbal Numerical Rating Scale (VNRS). This scale ranges from 0 to 10, with 0 being no pain and 10 being worst pain.
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lidocaine Treatment Group | Placebo Treatment Group
Number analyzed (Participants) | 16 | 12
units on a scale | -3.8 [-5.3 to -2.2] | -4.0 [-5.5 to -2.5]
Statistical Analysis 1: Comparison: Lidocaine Treatment Group vs Placebo Treatment Group; Outcome was residual change score calculated by regressing immediate postop pain on 24 hour pain. This allows patient to serve as own control for intial values; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-1.2 to 2.1]

2. Primary Outcome: Pain Change in 24 Hours (Self Reported Pain From Electronic Health Records)
Description: Pain will be measured by the Verbal Numerical Rating Scale (VNRS). This scale ranges from 0 to 10, with 0 being no pain and 10 being worst pain.
Time Frame: Immediate post-op to 24 hours post op
Population: This was an intention to treat analysis. Pain was measured with self reported pain from electronic health records and improvement was change from immediate post-op to 24 hours post-op (pain at 24 hours minus pain immediate postop) Assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lidocaine Treatment Group | Placebo Treatment Group
Number analyzed (Participants) | 16 | 12
units on a scale | -2.1 [-4.6 to -0.5] | -4.0 [-5.1 to -2.9]
Statistical Analysis 1: Comparison: Lidocaine Treatment Group vs Placebo Treatment Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-1.77 to 1.49], Standard Error of Mean 0.79

3. Secondary Outcome: Change in Hydromorphone in 24 Hours
Description: This was an intention to treat analysis. records and improvement was change from immediate post-op to 24 hours post-op (pain at 24 hours minus pain immediate postop) Assessment. Hydromorphone was quantified as morphine milligram equivelents (MME).
Time Frame: Immediate post-op to 24 hours post op
Population: This was an intention to treat analysis. records and improvement was change from immediate post-op to 24 hours post-op (pain at 24 hours minus pain immediate postop) Assessment. There were n=3 in lidocaine group with no medication doses reported.
Measure: Mean (95% Confidence Interval); unit: milligram morphine equivalents (MME)
Arm/Group | Lidocaine Treatment Group | Placebo Treatment Group
Number analyzed (Participants) | 13 | 12
milligram morphine equivalents (MME) | 0.4 [-0.4 to 1.3] | 4.7 [-3.4 to 12.9]
Statistical Analysis 1: Comparison: Lidocaine Treatment Group vs Placebo Treatment Group; Outcome was residual change score calculated by regressing immediate postop hydromorphone on 24 hour hydromorphone. This allows patient to serve as own control for intial values; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-9.62 to 6.09], Standard Error of Mean 3.61

ADVERSE EVENTS:
Time Frame: 21 days
Description: 1. All-Cause Mortality: The occurrence of death due to any cause.
  2. SAE: adverse events that result in: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect.
  3. Other (Not Including Serious) Adverse Events: Adverse events that are not Serious Adverse Events.
Arm/Group | Lidocaine Treatment Group | Placebo Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 5/16 | 2/12
Other Adverse Events (participants affected / at risk) | 5/16 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine Treatment Group (N=16) | Placebo Treatment Group (N=12)
Infection at donor site (Infections and infestations) | 5 (5) | 2 (2) — Infection at donor site
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine Treatment Group (N=16) | Placebo Treatment Group (N=12)
Acute lood loss Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Graft failure (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Wound breakdown (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Prolongation of hospitalization (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT02229578/Prot_SAP_000.pdf